CLINICAL TRIAL: NCT03402581
Title: The Effect of Different Videolaryngoscopes on Intubation Success in Obese Patients
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, associated professor, Ankara University
Other Study IDs: 18-925-16
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Difficult Airway, Videolaryngoscopes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- c-mac used for intubation: obese patients intubated with c-mac videolaryngoscope
  Interventions: Device: c-mac laryngoscope
- mc-grath used for intubation: obese patients intubated with mc-grath videolaryngoscope
  Interventions: Device: c-mac laryngoscope

INTERVENTIONS:
Device: c-mac laryngoscope — type of laryngoscopes
  Other Names: mc-grath laryngoscope

SUMMARY:
Obese patients may have difficulty in airway management.Patients who have body mass index > 35 are challenging patients for anesthesiologist. Short neck, more adipose tissue may be reasons for airway difficulty. Videolaryngoscopes are devices that ease the management of difficult airway.This study is designed to evaluate the differences and the effects of different laryngoscopes.

ELIGIBILITY:
Inclusion Criteria:

* body mass index> 35

Exclusion Criteria:

* emergency airway

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective surgery and have body mass index > 35
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-09-02 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
intubation difficulty | 1 minute
  the management of airway

SECONDARY OUTCOMES:
airway assesment | 1 minute
  evaluating the airway

CONTACTS AND LOCATIONS:
Overall Officials: CIGDEM YILDIRIMGUCLU, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No